CLINICAL TRIAL: NCT00325546
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Fixed-Dose (Rimonabant 20mg), Multi-National, Multicentre Study of Weight-Reducing Effect and Safety of Rimonabant in Obese Patients With or Without Comorbidities
Brief Title: Study of Weight-Reducing Effect and Safety of Rimonabant In Obesity in ASIA (RIO-ASIA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC6001
Record Dates: First submitted 2006-05-12; First posted 2006-05-15 (Estimated); Last update posted 2009-04-07 (Estimated); Status verified 2009-04

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity | interventions — Rimonabant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Rimonabant (SR141716)
Drug: Placebo

SUMMARY:
Primary : effect on weight loss and weight maintenance over 9 months when prescribed with a hypocaloric diet in obese patients.

Secondary : effect on HDL-Cholesterol, triglycerides, fasting-insulin, fasting glucose, waist circumference - safety and tolerability

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI)> 25 kg/m²

Exclusion Criteria:

* Absence of stable weight (variation < 5 kg) within three months prior to screening visit),
* Absence of effective contraceptive method for females of childbearing potential,
* Presence of treated or untreated type 1 or type 2 diabetes,
* Systolic blood pressure > 165 mm Hg and/or diastolic blood pressure > 105 mm Hg on 2 consecutive visits from the screening to the inclusion visit,
* Presence of secondary hypertension,
* Patients with conditions/concomitant diseases making them non evaluable for the primary efficacy endpoint (presence of any clinically significant endocrine disease according to the Investigator, obesity of known endocrine origin...)
* Presence of any severe medical or psychological condition or chronic conditions/infections that in the opinion of the Investigator would compromise the patient's safety or successful participation in the study,
* Presence of any clinically significant abnormality according to the Investigator on the ECG performed on the inclusion visit.
* Presence or history of cancer within the past five years with the exception of adequately treated localized basal cell skin cancer or in situ uterine cervical cancer.
* Related to previous or concomitant medications :

  * Drugs affecting weight (e.g., sibutramine, orlistat, herbal preparations, etc).
  * Antidiabetic drugs.
* Related to laboratory findings:

  * Positive test for hepatitis B surface antigen and/or hepatitis C antibody.
  * Abnormal TSH level (TSH > ULN or < LLN).
  * Positive urine pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 643 (Actual)
Dates: Start 2006-04; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Absolute change in weight from baseline to month 9

SECONDARY OUTCOMES:
HDL-Cholesterol, triglycerides, fasting-insulin, fasting glucose, waist circumference(physical examination, vital signs, ECG, laboratory tests, adverse events).

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (3):
- Sanofi-Aventis, Shanghai, China
- Sanofi-Aventis, Seoul, South Korea
- Sanofi-Aventis, Taipei, Taiwan